CLINICAL TRIAL: NCT02568813
Title: Epilepsy and Mood Regulation Disorders: a Prospective and Longitudinal Study in Children With Newly Diagnosed Epilepsy
Brief Title: Epilepsy and Mood Regulation Disorder in Children
Acronym: EPILETRE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2013-834
Record Dates: First submitted 2015-09-30; First posted 2015-10-06 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Epilepsy
Keywords: epilepsy; depression; mood disorder; anxiety; cyclothymia; Behavioral neuropsychiatric features
MeSH Terms: conditions — Epilepsy; Depression; Mood Disorders; Anxiety Disorders; Cyclothymic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Scales passation (Experimental)
  Interventions: Behavioral: Multiscore Depression Inventory for Children scale

INTERVENTIONS:
Behavioral: Multiscore Depression Inventory for Children scale
  Other Names: Revisited Children's Manifest Anxiety Scale; Kochman indicating a cyclothymia disorder Scale; Weschler Intelligence Scale for Children - 4th Edition

SUMMARY:
Epilepsy is a multifaceted disorder and a major public health problem. In addition to recurrent and unpredictable seizures, abnormalities in psychiatric status, cognition and social-adaptive behaviors are potential major sources of disability in children and adults with epilepsy disorders. Recent studies have unequivocally documented raised psychiatric comorbidities in children with epilepsy, particularly emotional regulation disorders such as depression and anxiety, as compared to both the general population and the children with other medical disorders, neurological and non-neurological. A prevalence of 12% to 35% has been reported, compared to 3-8% in the general population.

Major advances have begun to uncover the potential mediators of emotional regulation disorders and social comorbidities in epilepsy, but important gaps remain in the early detection, treatment and prevention of these disorders. A very small number of investigations have examined children with epilepsy at or near the time of diagnosis. This is a time during which the effects of chronic epilepsy, potential averse social effects of epilepsy, and other complicating aetiological effects are minimized.

Epilepsy syndromes provide a useful framework for considering the risk and type of emotional dysregulation comorbidities. But variability within and across syndromes needs to be taken into account thus requiring a strict phenotyping by specialists in the filed of pediatric epileptology. Retrospective studies, usually including patients with chronic epilepsies and suffering from a mixed spectrum of epilepsy syndromes introduce biases leading to rather disparate findings.

Are such disorders the result of common physiopathological mechanisms, which precede the development of the epilepsy? The link between an underlying brain disorder and psychiatric comorbidities has emerged in recent literature, with evidence based on studies in adults, suggesting bidirectional relations between epilepsy and neurobehavioural comorbidities. Emotional regulation disorders can follow the onset of epilepsy, but they can also precede it, thus serving as a possible risk factor. The clinical implication of such a bidirectional association is that neurobehavioural comorbidities might be present at diagnosis and even before epilepsy onset. There is a need for greater understanding of the causes of these conditions in younger people.

The degree to which specific epilepsy syndromes are associated with the relative risk of emotional dysregulation disorders in children with new- or recent-onset (within six months prior to enrolment) has rarely been comprehensively examined and represents the focus of the current investigation.

The investigators study will be based on a prospectively recruited cohort of 280 children/adolescents with recently diagnosed epilepsy. All participating centres dispose of the necessary competences for a precise diagnosis of the epilepsy syndromes and the tools for a per case appropriate aetiology screening. Following a first seizure children are usually first examined at hospital based emergency departments. Prompt referral to the epilepsy teams participating at the present study will significantly reduce the population biases and shortcuts encountered in studies that recruited patients with chronic epilepsy followed in tertiary care epilepsy units.

The investigators expect their results to provide a greater understanding of both the shared and the unique features of emotional regulation disorders, in relation to specific epilepsy categories defined on the basis of the underlying physiopathological mechanisms.

Such knowledge will also assist clinicians and families in the planning of both diagnosis and management resources.

ELIGIBILITY:
Inclusion Criteria:

* one of the following 3 epilepsy categories (focal structural epilepsy, with or without (MRI-negative) detectable cerebral lesion; focal idiopathic (genetic) epilepsy; generalized idiopathic (genetic) epilepsy).
* Onset of epilepsy within the 6 months from enrolment.
* Patients whose eventual antiepileptic drug treatments were not modified in the months preceding the neuropsychological and psychiatric evaluations.
* Patients who give their consent to participate in the study and whose legal guardians have agreed to sign the written consent form.

Exclusion Criteria:

* Patients younger than 5 years and 11 months or older than 15 years and 6 months.
* Patients with a diagnosis of epilepsy, other than the types defined above.
* Cognitive impairment, defined as a score of <70, based on WISC-IV verbal comprehension and perceptual reasoning scales.
* Children with a confirmed diagnosis of a psychiatric disorder, other than those studied.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2015-03-30 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of children with new- or recent-onset epilepsy with a pathological score in a least one of the 3 scales | 18 months
  The 3 scales are MDI-C ; R-CMAS and Kochman scale :
  * A standard score of >66 for MDI-C (Multiscore Depression Inventory for Children) indicating a depressive disorder;
  * A standard score of >60 or <40 for R-CMAS (Revisited Children's Manifest Anxiety Scale) indicating an anxiety disorder;
  * A score of >12 for Kochman indicating a cyclothymia disorder

SECONDARY OUTCOMES:
Correlate pathological scores obtained with the type of epilepsy | 18 months
  The same scoring system as for the primary end point will be used
  Type of epilepsy :
  * with or without (MRI-negative) detectable cerebral lesion;
  * focal idiopathic (genetic) epilepsy;
  * generalized idiopathic (genetic) epilepsy).
Correlate pathological scores with the progression of epilepsy disease | 18 months
  The same scoring system as for the primary end point will be used to evaluate the development, or progression, of emotional regulation disorders after 18 months of follow-up (constituted epilepsy);
  In each types of epilepsy, progression of the disease will be assessed by :
  * crises frequency
  * crises type

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme Mère Enfant, Bron, Rhône, France